CLINICAL TRIAL: NCT01060189
Title: Hemostatic Effects of Ulinastatin and Tranexamic Acid in Cardiac Surgery With Cardiopulmonary Bypass: A Pilot Study
Brief Title: Hemostatic Effects of Ulinastatin and Tranexamic Acid in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, SHI Jia, Associated Professor and Vice Chair of department of anesthesiology, Fuwai Hospital, NCCD, PUMC & CAMS, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UTI Pilot Study
Record Dates: First submitted 2010-01-28; First posted 2010-02-02 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Hemostasis
Keywords: ulinastatin; tranexamic acid; cardiac surgery procedures; hemostasis
MeSH Terms: interventions — urinastatin; Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ulinastatin (Experimental): 1,000,000 units of ulinastatin in 50ml solution before skin incision; 50ml saline solution after neutralization
  Interventions: Drug: Ulinastatin
- Tranexamic Acid (Experimental): 15mg/kg tranexamic acid in 50ml solution before skin incision; 15mg/kg tranexamic acid in 50ml solution after neutralization
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): 50ml saline solution before skin incision; 50ml saline solution after neutralization
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Ulinastatin
  Arms: Ulinastatin
Drug: Tranexamic Acid
  Arms: Tranexamic Acid
Drug: Saline Solution
  Arms: Placebo

SUMMARY:
Antifibrinolytic drugs are used to decrease perioperative bleeding and allogeneic transfusions. The extensively studied antifibrinolytic drug aprotinin is efficacious but expensive, and has been proved to link to higher risks of serious side effects including renal problems, myocardial events, and strokes in patients undergoing CABG. After the secession of aprotinin in 2007, a marked increase of blood loss and transfusions in cardiac surgery took place. An effective and secure hemostatic agent is badly needed. Ulinastatin, urinary trypsin inhibitor(UTI), is a secreted Kunitz-type protease inhibitor with a wide inhibition spectrum, including plasmin. Limited studies offered clues to its antifibrinolytic effect. Tranexamic acid has been applied for years with convinced efficacy and safety. The objective of the study is to evaluate the hemostatic effect of ulinastatin and tranexamic acid in cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Atrial or ventricular septum defect patients requiring cardiac surgery with CPB
* Rheumatic or recessive valvular patients requiring valvular repair or replacement with CPB
* Coronary artery disease patients requiring coronary revascularization surgery with CPB

Exclusion Criteria:

* Non-primary cardiac surgery
* Definite liver or renal dysfunction
* Disorder in coagulation function
* Allergy
* Pregnancy or lactation
* Disabled in spirit or law
* Fatal conditions such as tumour

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Postoperative blood loss | Postoperatively
  Defined as the total volume of chest drainage postoperatively

SECONDARY OUTCOMES:
Rate of reexploration for bleeding | Postoperatively
Rate of major bleeding | Perioperatively
  Major bleeding is defined according to the CURE study
Transfusion of allogeneic erythrocytes | Perioperatively
  Rate of exposure and volume of allogeneic erythrocytes transfused
Transfusion of fresh frozen plasma (FFP) | Perioperatively
  Rate of exposure and volume of FFP transfused
Transfusion of allogeneic platelets | Perioperatively
  Rate of exposure and volume of allogeneic platelets transfused
Length of stay in ICU and hospital postoperatively | Postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Lihuan Li, MD, Study Chair — Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC; Jia Shi, MD, Principal Investigator — Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC
Locations (1):
- Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang P, Lv H, Qi X, Xiao W, Xue Q, Zhang L, Li L, Shi J. Effect of ulinastatin on post-operative blood loss and allogeneic transfusion in patients receiving cardiac surgery with cardiopulmonary bypass: a prospective randomized controlled study with 10-year follow-up. J Cardiothorac Surg. 2020 May 14;15(1):98. doi: 10.1186/s13019-020-01144-9. PMID 32410683